CLINICAL TRIAL: NCT02143518
Title: Phase 1 Study of the Safety and Immunogenicity of Na-GST-1/Alhydrogel, With or Without a CpG ODN Adjuvant, in Healthy Adults
Brief Title: Safety and Immunogenicity Study of Na-GST-1 With or Without CpG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SVI-GST-03
Record Dates: First submitted 2014-05-14; First posted 2014-05-21 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm; Necator americanus; Hookworm; Hookworm Disease; Iron-deficiency anemia; Soil-transmitted helminth infection; Neglected Tropical Disease; Na-GST-1; CpG
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency; Neglected Diseases | interventions — CPG-oligonucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 µg Na-GST-1/Alhydrogel (Experimental): High Dose Na-GST-1/Alhydrogel® Only
  Interventions: Biological: Na-GST-1/Alhydrogel®
- 30 µg Na-GST-1/Alhydrogel + CpG 10104 (Experimental): Low Dose Na-GST-1/Alhydrogel® Plus 500 µg CpG 10104
  Interventions: Biological: Na-GST-1/Alhydrogel®; Biological: CpG 10104
- 100 µg Na-GST-1/Alhydrogel + CpG 10104 (Experimental): High Dose Na-GST-1/Alhydrogel® Plus 500 µg CpG 10104
  Interventions: Biological: Na-GST-1/Alhydrogel®; Biological: CpG 10104

INTERVENTIONS:
Biological: Na-GST-1/Alhydrogel® — The Na-GST-1 candidate vaccine contains the recombinant Na-GST-1 protein expressed by Pichia pastoris. Purified Na-GST-1 was subsequently adsorbed onto aluminum hydroxide gel (Alhydrogel®) and suspended in a solution containing 10% glucose and 10 mM imidazole. The final concentration of Na-GST-1 in the drug product is 0.1 mg/ml whereas that of Alhydrogel® is 0.8 mg/ml. Different doses of Na-GST-1 will be delivered by injecting different volumes of the 0.1 mg/ml Na-GST-1 preparation.
  Other Names: Na-GST-1; Necator americanus glutathione S-transferase-1
Biological: CpG 10104 — Unmethylated cytosine-guanine dinucleotides (CpGs) are found in bacterial DNA in the expected frequency predicted by random usage, whereas their occurrence is suppressed 4-fold in vertebrate DNA. In vertebrate DNA CpG motifs are also usually methylated. Bacterial CpG-DNA motifs are recognized by the human innate immune system via Toll-like Receptor-9 (TLR-9), a pathogen-associated molecular pattern (PAMP) receptor that is expressed, in particular, by antigen-presenting dendritic cells. Interactions between CpG-DNA and TLR9 rapidly activate antigen-presenting dendritic cells to upregulate co-stimulatory molecules and to produce Th1-polarizing cytokines such as interleukin-12 and interferon gamma. CpG 10104 is a short synthetic oligodeoxynucleotide of the following sequence: 5'-TCG TCG TTT CGT CGT TTT GTC GTT-3'.
  Other Names: Cytosine-phosphate-Guanine oligodeoxynucleotide; CpG ODN 101014; CpG ODN
  Arms: 100 µg Na-GST-1/Alhydrogel + CpG 10104; 30 µg Na-GST-1/Alhydrogel + CpG 10104

SUMMARY:
Na-GST-1 is a protein expressed during the adult stage of the hookworm life cycle that is thought to play a role in the parasite's degradation of host hemoglobin for use as an energy source. Vaccination with recombinant GST-1 has protected dogs and hamsters from infection in challenge studies. This study will evaluate the safety and immunogenicity of two formulations of Na-GST-1 in healthy adult volunteers when co-administered with the immunostimulant CpG 10104, a Toll-like Receptor-9 agonist.

DETAILED DESCRIPTION:
This is a Phase 1 randomized double-blind dose-escalation clinical trial in healthy hookworm-naïve adults conducted at the George Washington Medical Faculty Associates, Washington, DC, and the George Washington University School of Medicine and Health Sciences, Department of Microbiology, Immunology and Tropical Medicine, Washington, DC. In total, 24 subjects will be progressively enrolled into 2 cohorts of 12 subjects each. In the first cohort 8 subjects will receive 30µg Na-GST-1/Alhydrogel co-administered with 500µg CpG 10104 and 4 subjects will receive 100µg Na-GST-1/Alhydrogel® only, in a randomized, double-blinded fashion. In the second cohort 8 subjects will receive 100µg Na-GST-1/Alhydrogel co-administered with 500µg CpG 10104 and 4 volunteers will receive 100µg Na-GST-1/Alhydrogel only, in a randomized, double-blinded fashion. Vaccinations will be administered intramuscularly in the deltoid muscle according to a 0, 2, 4-month schedule. Each subject will participate in the study for 68 weeks (16 months) and the total duration of the study is estimated at approximately 19 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 50 years, inclusive.
* Good general health as determined by means of the screening procedure.
* Available for the duration of the trial (68 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Able to understand and comply with planned study procedures.

Exclusion Criteria:

* Pregnancy as determined by a positive urine human choriogonadotropin (hCG) test (if female).
* Participant unwilling to use reliable contraception up until one month following the third immunization (if female and not surgically sterile, abstinent, at least 2 years post-menopausal, or determined otherwise by medical evaluation to be sterile).
* Currently lactating and breast-feeding (if female).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies. A history of essential hypertension that is well controlled by medication will not be considered exclusionary.
* Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing with the exception of greater than 1+ blood detected in females during menses).
* Laboratory evidence of hematologic disease (hemoglobin <11.1 g/dl [females] or <12.5 g/dl [males]; absolute leukocyte count <3400/mm3 or >10.8 x 103/mm3; or platelet count <140,000/mm3).
* Laboratory evidence of a coagulopathy (activated PTT or PT INR greater than 1.1-times the upper reference limit).
* Serum glucose greater than 1.2-times the upper reference limit.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Planned participation in another investigational vaccine or drug trial within 30 days of starting this study or until Visit #17 (6 months after the third vaccination).
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for daily use of inhalers, or emergency clinic visit or hospitalization within 6 months of the volunteer's expected first vaccination in the study.
* Positive test for hepatitis B surface antigen (HBsAg).
* Positive confirmatory test for HIV infection.
* Positive confirmatory test for hepatitis C virus (HCV) infection.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of the volunteer's expected first vaccination in this study or planned use up to one month following the last vaccination.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to the volunteer's expected first vaccination in the study.
* Previous receipt of the Na-GST-1/Alhydrogel® hookworm vaccine.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosis, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia; or laboratory evidence of possible autoimmune disease determined by a positive anti-dsDNA titer, positive rheumatoid factor, proteinuria and/or a positive ANA.
* History of previous infection with hookworm or residence for more than 6 months in a community where hookworm is endemic.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- Available data/document: Clinical Study Report — https://gwvru.smhs.gwu.edu/clinical

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 100 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel + CpG 10104
Started | 8 | 8 | 8
Completed | 8 | 6 | 7
Not Completed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel + CpG 10104 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.5 [24.75 to 30.5] | 31.0 [26.0 to 45] | 32 [28.5 to 41.75] | 29 [25.5 to 41.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 10
  Male | 3 | 6 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 5 | 4 | 10
  White | 5 | 1 | 4 | 10
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Vaccine-related Adverse Events
Description: The frequency of immediate, systemic, and local injection site adverse events, graded by severity, for Na-GST-1/Alhydrogel administered alone or in combination with CpG 10104
Time Frame: Up to study day 470
Measure: Count of Participants; unit: Participants
Arm/Group | 100 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel + CpG 10104
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Number of participants with an immediate AE | 1 | 3 | 0
  Number of participants with a systemic AE | 3 | 4 | 5
  Number of participants with an injection site AE | 7 | 8 | 7

2. Secondary Outcome: IgG Antibody Response to Na-GST-1 on Study Day 126
Description: Dose and formulation of Na-GST-1 that generates the highest IgG antibody response at Day 126 (14 days after final vaccination), as determined by a qualified indirect enzyme-linked immunosorbent assay (ELISA) and measured in Arbitrary Units (AU) that are interpolated from a standard reference curve formulated by serial dilutions of a serum pool derived from known high responders in previous clinical trials of this antigen. This ELISA has not been validated and does not report mass units since these have not yet been defined. Reporting ELISA values in AU is an accepted practice early in clinical development before full assay validation and quantification of mass units.
Time Frame: 14 days after final vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Arbitrary Units/mL
Arm/Group | 100 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel + CpG 10104
Number analyzed (Participants) | 8 | 6 | 7
Arbitrary Units/mL | 49.42 [17.07 to 143.0] | 300.7 [194.6 to 464.8] | 389.5 [212.8 to 713.0]

3. Secondary Outcome: Exploratory Cellular Immune Response to Na-GST-1
Description: Exploratory studies of the cellular immune responses to the Na-GST-1 antigen both before and after immunization.
Time Frame: Up to study day 290
Population: The data for this endpoint were not collected since PBMC samples were not sent from the clinical trial site in Africa to the testing laboratory in the US due to the ending of the grant funding the study and a lack of funding to ship the samples. This endpoint will not be completed.
Arm/Group | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel | 100 µg Na-GST-1/Alhydrogel + CpG 10104
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for approximately 68 weeks, or 16 months. This includes following participants for approximately 12 months after receiving the third vaccination.
Arm/Group | 100 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel + CpG 10104 | 100 µg Na-GST-1/Alhydrogel + CpG 10104
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 µg Na-GST-1/Alhydrogel (N=8) | 30 µg Na-GST-1/Alhydrogel + CpG 10104 (N=8) | 100 µg Na-GST-1/Alhydrogel + CpG 10104 (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Antinuclear antibody increased (Investigations) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Body temperature increased (Investigations) | 1 | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Diastolic hypertension (Vascular disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3
Haemoglobin decreased (Investigations) | 2 | 1 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hangover (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 1
Injection site coldness (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 1 | 1 | 0
Injection site pain (General disorders) | 7 | 8 | 7
Injection site pruritus (General disorders) | 1 | 0 | 0
Injection site swelling (General disorders) | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 3 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 6
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Vaginitis bacterial (Infections and infestations) | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No